CLINICAL TRIAL: NCT01363349
Title: A Randomized, Double-Blind, Active-Controlled,Phase 2/3 Study to Determine the Short-Term (6-Week) and Long-Term (6 Month) Cognitive and Anti-Psychotic Efficacy, Safety and Tolerability of CYP-1020 Compared to Risperidone in Patients With Schizophrenia
Brief Title: Phase IIb-III Study of BL-1020 Small Molecule for Schizophrenia
Acronym: CLARITY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: pre-planned interim analysis of the Phase II/III CLARITY trial of BL-1020 indicate that the trial would not meet the pre-specified primary efficacy endpoint.
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1020-CLIN-201; NCT01365299 (obsolete NCT alias)
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia; Cognitive Effect on Schizophrenic Patients
MeSH Terms: conditions — Schizophrenia | interventions — perphenazine GABA ester; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYP-1020 (Experimental): Dose titration 15-35mg/day for 6 months
  Interventions: Drug: CYP-1020
- Risperidone (Active Comparator): Dose titration 2-6mg/day for 6 months
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: CYP-1020 — CYP-1020 (formerly known as BL-1020) is an orally available new chemical entity.
  Other Names: BL-1020
  Arms: CYP-1020
Drug: Risperidone
  Arms: Risperidone

SUMMARY:
This is a randomized, double-blind, active-controlled, 6 month study designed to evaluate the cognitive effects of treatment with CYP-1020 compared to risperidone. The primary efficacy endpoint will occur after 6 weeks of treatment; additional (secondary) efficacy endpoints will occur after 12 and 24 weeks of treatment.

Up to 450 patients will be randomized to CYP-1020 or risperidone in a 1:1 ratio. The study will utilize a flexible dose escalation scheme designed to allow patients to titrate to their maximally tolerated dose; doses of CYP-1020 may range from a minimum of 15 mg to a maximum of 35 mg, whereas doses of risperidone will range from a minimum of 1 mg to 3 mg BID (2-6 mg daily). To ensure effective blinding across all treatment groups, all patients will be treated twice daily with study drug and/or placebo, as indicated (i.e., double-dummy design).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant or lactating female, 18-50 years of age inclusive
2. Patients must have exhibited symptoms meeting the criteria of schizophrenia for at least one year, but not more than 20 years, prior to Screening
3. Recent onset (not more than 30 days) of worsening of psychiatric symptoms at Screening.
4. Currently experiencing an acute exacerbation of schizophrenia, as defined by the following results at Screening and Baseline:

   * ≥70 total score on the PANSS
   * ≥4 (moderate) on two of the following four PANSS items: (1) delusions, (2) hallucinatory behaviors, (3) conceptual disorganization or (4) suspiciousness/persecution, where at least one of the two items must be either delusions or hallucinatory behaviors
5. CGI-S score between 4 and 6 (moderately ill to severely ill) at the Screening and Baseline visits.
6. Has exhibited a sufficient clinical response to at least one previous course of an anti-psychotic agent prescribed at a generally recognized therapeutic dose.
7. Must have completed at least 5 years of formal education or its equivalent

Exclusion Criteria:

1. Breastfeeding or pregnant
2. Symptoms of schizophrenia for more than 20 years at the time of screening.
3. Psychotic symptoms that have failed to improve (based on Investigator's opinion or documented medical history) following sufficient treatment with therapeutic doses of two or more anti-psychotics agents over the preceding 2 years
4. Prior history of neuroleptic malignant syndrome
5. Prior history or current evidence of moderate or severe tardive dyskinesia (mild is acceptable).
6. Abnormal ECG evaluation
7. History of confirmed epilepsy or prior seizure disorder (history of a single febrile seizure is not exclusionary)
8. In the opinion of the investigator, unstable medical disease (e.g., malignancy, poorly controlled diabetes or hypertension, ischemic cardiac disease, dilated cardiomyopathy or valvular heart disease, pulmonary disease, liver disease, kidney disease)
9. Acute infectious disease (e.g., malaria, dengue fever, hepatitis A), or chronic infectious disease (e.g., history of AIDS or HIV positivity, tuberculosis)
10. Likely allergy, sensitivity or intolerance to BL-1020, perphenazine, risperidone, paliperidone, or any of the drug product excipients
11. Any suicide attempt within the preceding 2 years
12. Any Substance Dependence disorder
13. High likelihood of substance abuse
14. Diagnosis with one of the following DSM-IV-TR Axis I diagnoses: schizophreniform disorder, schizoaffective disorder, bipolar disorder, substance dependency, mood disorder with psychotic features; psychotic disorder NOS
15. Requiring chronic treatment with benzodiazepines
16. Requiring chronic treatment with mood stabilizers
17. Previously treated with clozapine within 6 months prior to screening
18. Any abnormal clinical laboratory test result that is judged by the Investigator to be clinically significant
19. History of, or serologic evidence of, acute or chronic active hepatitis B or C

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 269 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Aharon, MD, Study Chair — BioLineRx, Ltd.
Locations (39):
- India (18):
  - Department of Psychiatry, Sheath VS General Hospital, Sheath KM School of Post Graduate Medicine & Research, Ahmedabad
  - Saoji Tupkari Hospital, Aurangabad
  - Spandana Nursing Home, Bangalore
  - KHM Hospital, Chennai
  - Asha Hospital, Hyderabad
  - Department of Psychiatry, Owaisi Hospital & Research Centre, Hyderabad
  - RK Yadav Memorial Mental Health and De-addiction Hospital, Jaipur
  - Mahendru Psychiatric Centre, Kanpur
  - Dreamland Nursing Home, Kolkata
  - Dayanand Medical College & Hospital, Ludhiana
  - Centre for Psychiatric Research, Department of Psychiatry, K.S Hegde Medical Academy, Mangalore
  - Jaslok Hospital&Research Centre, Mumbai
  - JSS Medical College Hospital, Mysore
  - Sujata Birla Hospital, Nashik
  - Vimhans Hospital, New Delhi
  - S.V.Medical College, Tirupati
  - Deva Mental Health Care, Varanasi
  - Vijayawada Institute of Mental Health & Neurosciences, Vijayawada
- Moldova (3):
  - IMSP Spitalul Clinic de Psihiatrie, Sectia 14, Chisinau
  - IMSP Spitalul Clinic de Psihiatrie, Sectia 17, Chisinau
  - IMSP Spitalul Clinic de Psihiatrie, Sectia 8, Chisinau
- Romania (18):
  - pitalul Clinic Judetean de Urgenta Arad Clinica Psihiatrie, Arad
  - Spitalul de Psihiatrie si Neurologie Brasov, Brasov
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Al. Obregia", Bucharest
  - Spitalul Clinic de Psihiatrie Dr. Alexandru Obregia Department 13, Bucharest
  - Spitalul Clinic de Psihiatrie Dr. Alexandru Obregia Department 1, Bucharest
  - Spitalul Clinic de Psihiatrie Dr. Alexandru Obregia Department 8, Bucharest
  - Spitalul Clinic de Psihiatrie Dr. Alexandru Obregia Department 9, Bucharest
  - Spitalul de Psihiatrie C.E.T.T.T. "Sf. Stelian", Bucharest
  - Spitalul Judetean Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Constanţa Clinica de Psihiatrie, Constanța
  - Spitalul Clinic de Neuropsihiatrie Clinica de Psihiatrie nr. 2, Craiova
  - Spitalul de Neuropsihiatrie Clinica de Psihiatrie I, Craiova
  - Spitalul Clinic de Psihiatrie Socola, Iași
  - Spital Clinic de Neurologie si Psihiatrie Oradea, Oradea
  - Spitalul Clinic Municipal "Dr.Gavril Curteanu" Oradea, Oradea
  - Spitalul de Psihiatrie "Dr. Gh. Preda", Sibiu
  - Spitalul Judetean de Urgenta Targoviste Clinica Psihiatrie Adulti nr. 7, Târgovişte
  - Spitalul Clinic Judetean Mures, Clinica Psihiatrie Nr. 2, Târgu Mureş

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone: 2-6 mg, 6 months
  Risperidone
Period: Overall Study
Arm/Group | CYP-1020 | Risperidone
Started | 133 | 136
Randomized | 133 | 136
Completed | 66 | 66
Not Completed | 67 | 70
Not completed — Adverse Event | 6 | 7
Not completed — Lack of Efficacy | 3 | 10
Not completed — Non compliance/Protocol deviations | 2 | 2
Not completed — Withdrawal by Subject | 14 | 6
Not completed — Lost to Follow-up | 5 | 6
Not completed — Not reported | 36 | 37
Not completed — missing | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP-1020 | Risperidone | Total
Number analyzed (Participants) | 133 | 136 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (8.76) | 32.3 (7.97) | 32.8 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 84 | 87 | 171
Race/Ethnicity, Customized [Number; unit: number of participants]
  asian | 92 | 94 | 186
  caucasian | 41 | 42 | 83
Region of Enrollment [Number; unit: participants]
  Romania | 41 | 42 | 83
  India | 92 | 94 | 186

OUTCOME MEASURES:

1. Primary Outcome: Cognition
Description: To evaluate the cognitive benefits of treatment with CYP-1020 (formerly known as BL-1020) compared to risperidone after 6 weeks of treatment in patients experiencing acute exacerbation of schizophrenia. Assessed by calculating difference between CYP-1020 and Risperidone on mean change from baseline to Week 6 endpoint on MATRICS Consensus Cognition Battery (MCCB) normative composite score. MCCB is a neuropsychological test battery that comprises 10 measures of 7 different cognitive areas including speed of processing, verbal learning, memory-verbal and non verbal reasoning and problem solving, visual learning, social cognition, attention/vigilance.The study was terminated after the interim analysis. MCBB total score ranges from -50 to 150. Change from Baseline by Visit (LOCF)Higher score means better cognitive functioning.
Time Frame: Baseline and 6 weeks
Population: Analysis for MCCB Score ITT population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CYP-1020 | Risperidone
Number analyzed (Participants) | 133 | 136
Scores on a scale
  MCCB Baseline Score | 8.7 (13.66) | 8.2 (13.86)
  MCCB Week 6 Score | 13.5 (12.92) | 12.5 (13.68)

2. Secondary Outcome: Long Term Cognition
Description: Evaluation of the cognitive benefits of treatment with BL-1020 compared to risperidone after 12 and 24 weeks of treatment
Time Frame: 12 and 24 weeks of treatment

3. Secondary Outcome: Long Term Schizophrenia Treatment
Description: Evaluation of the antipsychotic efficacy of BL-1020 compared to risperidone after 6, 12 and 24 weeks of treatment
Time Frame: Baseline and 6, 12 and 24 weeks of treatment

ADVERSE EVENTS:
Arm/Group | CYP-1020 | Risperidone
Serious Adverse Events (participants affected / at risk) | 6/133 | 5/136
Other Adverse Events (participants affected / at risk) | 105/133 | 101/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP-1020 (N=133) | Risperidone (N=136)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
schizophrenia (Psychiatric disorders) | 2 (2) | 3 (3)
completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
delerium (Psychiatric disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
persecutory delusion (Psychiatric disorders) | 1 (1) | 0 (0)
sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP-1020 (N=133) | Risperidone (N=136)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 32 (32) | 24 (24)
TREMOR (Nervous system disorders) | 30 (30) | 28 (28)
AKATHISIA (Nervous system disorders) | 18 (18) | 18 (18)
SOMNOLENCE (Nervous system disorders) | 11 (11) | 12 (12)
SEDATION (Nervous system disorders) | 8 (8) | 2 (2)
INSOMNIA (Psychiatric disorders) | 20 (20) | 26 (26)
RESTLESSNESS (Psychiatric disorders) | 11 (11) | 12 (12)
ANXIETY (Psychiatric disorders) | 8 (8) | 9 (9)
vomiting (Gastrointestinal disorders) | 8 (8) | 3 (3)
salivary hypersecretion (Gastrointestinal disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No